CLINICAL TRIAL: NCT06167486
Title: A Phase I Clinical Study to Evaluate the Safety Tolerability and Preliminary Efficacy of SG2918 in Subjects With Advanced Malignant Tumors
Brief Title: SG2918 For Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-2918-101
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG2918 (Experimental): SG2918 monotherapy
  Interventions: Drug: SG2918

INTERVENTIONS:
Drug: SG2918 — The SG2918 will be administrated by intravenous infusion every 3 weeks

SUMMARY:
This is a Phase I, open-label, dose escalation and dose expansion study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SG2918 in subjects with Advanced Malignant Tumors who are refractory or resistant to standard therapy, or without available standard or curative therapy.

DETAILED DESCRIPTION:
The study consists of dose escalation and dose expansion, the dose escalation will be performed in a standard 3+3 manner at the dose of 0.1mg/kg、0.5mg/kg、1 mg/kg、1.5mg/kg、2 mg/kg、2.5mg/kg and 3 mg/kg, and the dose expansion will be done in specific tumor types. Patients enrolled in the study will receive SG2918 treatment every three weeks (Q3W), until disease progression, intolerable toxicity or others, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented advanced malignant tumors that is refractory/relapsed to standard therapies;
2. Adequate organ function;
3. ECOG Performance Status score of 0 or 1;
4. Must have at least one measurable lesion according to RECIST Version1.1;
5. Toxicity caused by prior anti-tumor therapy recovered to Grade 0 to 1 (CTCAE 5.0);
6. Must have an effective contraception during the study, starting with the Screening Visit through 7 months after the last dose of study intervention.

Exclusion Criteria:

1. Has active central nervous system metastatic lesions;
2. Has Active autoimmune disease requiring systemic therapy within the past 2 years;
3. Has Grade 2 and above peripheral neuropathy;
4. Has an active infection requiring systemic therapy;
5. Has a history of any of the following cardiovascular conditions within 6 months of dosing: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, coronary artery bypass graft, pulmonary embolism, etc; has New York Heart Association (NYHA) Class II and above congestive heart failure; LVEF<50%;
6. Has a history of hypertensive crisis or hypertensive encephalopathy; Uncontrolled hypertension though standard treatment within 14 days before the first dose (systolic blood pressure≥160 mmHg and/or diastolic blood pressure≥100mmHg);
7. Has known human immunodeficiency virus (HIV) and/or hepatitis B or C infections;
8. Has a history of potent CYP3A4 inhibitor with 2 weeks;
9. Has received systemic anticancer therapy, radiotherapy, or surgery within 4 weeks before the start of study treatment;
10. Have received previous treatment targeted LILRB4 or MMAE experiencing serious adverse events;
11. Have received previous immunotherapy experiencing serious adverse events that leading to permanent discontinuation;
12. Have received systemic corticosteroids (equivalent dose > 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to the first dose;
13. Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody (mAB) and or any components of the study intervention;
14. Any live vaccine within 28 days prior to the first dose;
15. Has a history of interstitial lung disease or active pneumonia or tracheal fistula; uncontrolled pleural, abdominal and pericardial effusion;
16. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the time of first dose until 30 days after last dose of SG2918
  Number and percentage of AEs which is calculated by worst CTCAE grade by CTCAE 5.0
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | Cycle 1 (up to 21 days)
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria and assessed as related to study drug, and unrelated to disease, disease progression, intercurrent illness or concomitant medications that occurs within the first cycle (three weeks) of treatment.

SECONDARY OUTCOMES:
Pharmacokinetics(PK): Cmax | From the time of first dose until 30 days after last dose of SG2918
  Maximum drug concentration after administration
Pharmacokinetics (PK): AUC | From the time of first dose until 30 days after last dose of SG2918
  Area Under the Curve of the drug after administration
Pharmacokinetics (PK): T1/2 | From the time of first dose until 30 days after last dose of SG2918
  Elimination half-life of the drug after administration
Pharmacokinetics (PK): CL | From the time of first dose until 30 days after last dose of SG2918
  Clearance of the drug after administration
Pharmacodynamic(PD): cellular biomarkers | From the time of first dose until 30 days after last dose of SG2918
  cellular biomarkers including CD4+ T cells, CD8+ T cells, Myeloid-derived suppressor cells (MDSCs) and Regulatory T cells (Tregs)
Pharmacodynamic(PD): cytokine levels | From the time of first dose until 30 days after last dose of SG2918
  Peripheral blood cytokine levels including measurements for TNF-α，IFN-γ，IL-2，IL-4、IL-6，IL-8，IL-10，IL-1β
Immunogenicity endpoints | Through study completion, an average of one year，assessed up to approximately 12 months
  Levels of anti-drug antibodies(ADAs) and neutralizing antibodies (tested in ADA-positive samples)
Efficacy endpoints | Through study completion, an average of one year，assessed up to approximately 12 months
  objective response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai first maternity and infant hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No